CLINICAL TRIAL: NCT06060665
Title: IDEAL: A 52-week, Double-blind, Placebo-controlled, Randomized, Phase 3 Study Intended to Determine the Effects of Seladelpar on Normalization of Alkaline Phosphatase Levels in Subjects With Primary Biliary Cholangitis (PBC) and an Incomplete Response or Intolerance to Ursodeoxycholic Acid (UDCA)
Brief Title: Intended to Determine the Effects of Seladelpar on Normalization of Alkaline Phosphatase Levels in Subjects With Primary Biliary Cholangitis (PBC)
Acronym: IDEAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB8025-32251; 2024-517409-10-00 (EU CTIS Number)
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2025-05-05 (Actual); Status verified 2025-05

CONDITIONS: Primary Biliary Cholangitis
Keywords: Primary Biliary Cholangitis (PBC); PBC
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — seladelpar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Seladelpar (Experimental): Participants will receive Seladelpar 10 mg one capsule daily for up to 52 weeks.
  Interventions: Drug: Seladelpar 10 mg
- Placebo (Experimental): Participants will receive placebo-to-match one capsule daily for up to 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Seladelpar 10 mg — Administered orally
  Arms: Seladelpar
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
To Determine the Effects of Seladelpar on Normalization of Alkaline Phosphatase Levels in Subjects with Primary Biliary Cholangitis (PBC) and an Incomplete Response or Intolerance to Ursodeoxycholic Acid (UDCA).

The primary objective is to evaluate the effect of seladelpar treatment at Week 52 compared to placebo based on normalization of alkaline phosphatase (ALP) defined by a composite endpoint of ALP ≤ 1.0× upper limit of normal (ULN) and ≥ 15% decrease from baseline in PBC participants with an ALP value greater than ULN but less than 1.67× ULN.

ELIGIBILITY:
Key Inclusion Criteria:

Individuals must meet the following criteria to be eligible for study participation:

1. Male or female with a diagnosis of primary biliary cholangitis (PBC) based on history.
2. Ursodeoxycholic acid (UDCA) for the 12 months prior to screening (with stable dose for > 3 months prior to screening) OR intolerant to UDCA (last dose of UDCA > 3 months prior to screening).
3. ALP > 1× ULN and < 1.67× ULN.
4. Females of reproductive potential must use at least 1 barrier contraceptive and a second effective birth control method during the study and for at least 90 days after the last dose. Male participants who are sexually active with female partners of reproductive potential must use barrier contraception, and their female partners must use a second effective birth control method during the study and for at least 90 days after the last dose.

Key Exclusion Criteria:

1. Previous exposure to seladelpar (MBX-8025).
2. A medical condition other than PBC that, in the Investigator's opinion, would preclude full participation in the study (eg, cancer) or confound its results.
3. Advanced PBC as defined by the Rotterdam criteria.
4. Laboratory parameters measured by the Central Laboratory at screening.
5. Clinically important hepatic decompensation.
6. Other chronic liver diseases.
7. Known history of human immunodeficiency virus (HIV) or positive antibody test at screening.
8. Clinically important alcohol consumption, defined as more than 2 drink units per day in women and 3 drink units per day in men, or inability to quantify alcohol intake reliably.
9. History of malignancy diagnosed or treated, active or within 2 years, or ongoing evaluation for malignancy; localized treatment of squamous or noninvasive basal cell skin cancers and cervical carcinoma in situ is allowed if appropriately treated prior to screening.
10. History of drug abuse that would compromise the quality of the clinical study.
11. Treatment with obeticholic acid or fibrates 6 weeks prior to screening.
12. Treatment with colchicine, methotrexate, azathioprine, or long-term systemic corticosteroids within 2 months prior to screening.
13. Initiation or dose adjustment of anti-pruritic drugs indicated for the treatment of pruritus within 1 month prior to screening.
14. Immunosuppressant therapies within 6 months prior to screening.
15. Other medications that affect liver or gastrointestinal functions, as well as the roux-en-y gastric bypass procedure, may be prohibited and should be discussed with the medical monitor on a case by-case basis.
16. Treatment with any other investigational therapy or device within 30 days or within halflives, whichever is longer, prior to screening.
17. Pregnancy or plans to become pregnant, or breastfeeding.
18. Any other condition(s) that would compromise the safety of the individual or compromise the quality of the clinical study, as judged by the investigator.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Response defined as Alkaline phosphatase (ALP) ≤ 1.0× Upper Limit of Normal (ULN) AND ≥ 15% Decrease in ALP at Week 52. | 52 weeks
Type, Frequency, and Severity of Treatment-emergent Adverse Events. | 52 weeks

SECONDARY OUTCOMES:
Percentage of Participant Response Defined as ALP ≤ 1.0× ULN. | 52 weeks
Percentage of Participant Response Defined as ALP ≤ 1.0× ULN AND ≥ 15% Decrease in ALP at 4 Weeks. | 4 weeks
Percentage of Participant Response Defined as ALP ≤ 1.0× ULN AND ≥ 15% Decrease in ALP at 12 Weeks. | 12 weeks
Percentage of Participant Response Defined as ALP ≤ 1.0× ULN AND ≥ 15% Decrease in ALP at 26 Weeks. | 26 weeks
Percentage of Participant Response Defined as ALP ≤ 1.0× ULN AND ≥ 15% Decrease in ALP at 39 Weeks. | 39 weeks
Absolute and Percent Change From Baseline in ALP. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (45):
- United States (43):
  - The Institute for Liver Health II LLC dba Arizona Clinical Trials; Arizona Liver Health, Chandler, Arizona
  - California Liver Research Institute, Pasadena, California
  - University of California (UC) Davis Medical Center, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado Denver - School of Medicine - Anschutz Medical Campus, Aurora, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Florida Research Institute, Lakewood Rch, Florida
  - University of Miami - Schiff Center for Liver Diseases, Miami, Florida
  - Gastro Health Research, Miami, Florida
  - Covenant Metabolic Specialists, LLC, Sarasota, Florida
  - Covenant Metabolic Specialists, LLC, Tampa, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Northwestern Medicine Clinical Research Unit (CRU), Chicago, Illinois
  - Tulane University Medical Center, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center - Baltimore, Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Kansas City Research Institute, Kansas City, Missouri
  - New-York-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Northwell Health Center for Liver Disease and Transplantation, Manhasset, New York
  - New York University (NYU) Langone Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of Rochester Medical Center - Strong Memorial Hospital, Rochester, New York
  - Gastro Health Research, Liberty Township, Ohio
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Center for Liver Health, Pittsburgh, Pennsylvania
  - OGI - Gastro One, Cordova, Tennessee
  - Galen Hepatology, Hixson, Tennessee
  - Gastrointestinal Associates of Northeast Tennessee, P.C., Johnson City, Tennessee
  - American Research Corporation - San Antonio, TX, Austin, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Liver Center of Texas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Soma Clinical Trials, LLC, Denison, Texas
  - Baylor College of Medicine - Baylor Clinic, Houston, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - Bon Secours Liver Institute of Hampton Roads, Richmond, Virginia
  - Velocity Clinical Research - Seattle, Seattle, Washington
  - Stanford University, Seattle, Washington
- Canada (2):
  - Centre de Recherche du Centre Hospitallier de I'Universite de Montreal (CRCHUM), Montreal
  - (G.I.R.I.) GI Research Institute Foundation, Vancouver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06060665